CLINICAL TRIAL: NCT01538524
Title: Analysis of Patient Seeking Second Opinion Who Undergoing Full Mouth Orthodontic Treatment
Brief Title: Analysis of Patient Seeking Second Opinion Who Are Undergoing Full Mouth Orthodontic Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201109008RB
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-01

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patient safety is a great concern for the whole society. Since the investigators have a leadership in the medical field in Taiwan, the investigators should be courageous to face the reality from the patients seeking second opinions undergoing orthodontic treatment.

Orthodontics just became a recognized specialty by the Department of Health in Taiwan in 2009. It is just a beginning to set up the training course criteria at the national level. It will be a good timing for us to look at the treatment quality when patients seeking second opinions at NTUH. Whether the unsatisfied results are from the patient's unrealistic expectation, patient's compliance issue, doctor's diagnosis, treatment planning or skills, or a simple communication problem, depend on a good systemic analysis from the records and questionnaire collected in a timely fashion.

The investigators plan to ask patients who are undergoing full-mouth orthodontic treatment and seeking second opinion to join this study. The investigators will thoroughly explain to patients before they agree to take records and fill in questionnaire. Then the investigators use these records to perform root cause analysis.

Our hypothesis is that the risk of adverse event (AE) is related to the training quality, communication skills, patient's understanding and compliance. From these results, the investigators shall be able to assess the risk of AE and make the education policy either at continued education level or special training courses towards a patient satisfied treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are not under full mouth fixed orthodontic treatment in National Taiwan University Hospital

Exclusion Criteria:

* Patient who only had partial orthodontic treatment
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are not under full mouth fixed orthodontic treatment in National Taiwan University Hospital
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-02; Study Completion 2014-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pi-Huei Liu, Principal Investigator — National Taiwan University Hospital